CLINICAL TRIAL: NCT00199550
Title: A Prospective Randomized Clinical Trial of Bipolar vs Monopolar Transurethral Resection of the Prostate (TURP)
Brief Title: Bipolar vs Monopolar Transurethral Resection of the Prostate (TURP)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Gyrus ACMI, Inc. (Other)
Responsible Party: Dr. Hassan Razvi, The University of Western Ontario
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R-04-533
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2008-07-29 (Estimated); Status verified 2008-07

CONDITIONS: BPH; Benign Prostatic Hyperplasia
Keywords: Transurethral Resection of Prostate; TURP
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (Active Comparator): Bipolar Electrosurgical Unit
  Interventions: Procedure: Bipolar Transurethral Resection of the Prostate
- 1 (Active Comparator): Monopolar Electrosurgical Unit
  Interventions: Procedure: Monopolar Transurethral Resection of the Prostate

INTERVENTIONS:
Procedure: Bipolar Transurethral Resection of the Prostate — Bipolar TURP
  Other Names: Vista, Bipolar TURP
  Arms: 2
Procedure: Monopolar Transurethral Resection of the Prostate — Monopolar TURP
  Other Names: Monopolar TURP
  Arms: 1

SUMMARY:
This study will prospectively evaluate a new electrosurgical procedure (bipolar transurethral prostatectomy) in men with symptomatic benign prostatic hyperplasia.

DETAILED DESCRIPTION:
The purpose of this study is to demonstrate that the Bipolar TURP using the Vista Controlled Tissue Resection System is safe and efficacious as a surgical treatment for men with symptomatic BPH, allowing a reduction in the post-operative hospitalization. It is expected that bipolar TURP will be safe and efficacious for the surgical treatment of BPH and will allow a < 24 hour post-operative hospital stay in > 50% of patients undergoing this procedure.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic benign prostatic hyperplasia including patients with acute urinary retention;
* Peak urinary flow rate < 12 ml/sec;
* American Urological Association (AUA) symptom score > 12.

Exclusion Criteria:

* Previous open or transurethral prostatic surgery;
* History of urethral stricture;
* Failure to discontinue alpha-adrenergic blocking agents for at least 14 days prior to surgery;
* Failure to discontinue 5-alpha reductase inhibitor for at least 1 month prior to surgery;
* Patient interested in future fertility;
* Patient with known neurogenic bladder dysfunction;
* Untreated urinary tract infection;
* American Society of Anesthesiologist (ASA) Class >III;
* Patients requiring anticoagulation with Coumadin or Heparin;
* Patient unable or unwilling to comply with follow-up schedule.

Ages: 50 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2004-05; Primary Completion 2008-03 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Evaluation of efficacy will be determined by comparing pre and post-operative symptom scores. | 6 months

SECONDARY OUTCOMES:
Pre and post-operative objective and subjective data for each treatment group will be assessed to determine safety and efficacy. Complications related to the surgical procedure will be noted by flexible cystoscopy at 6 months. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Hassan Razvi, MD, FRCSC, Principal Investigator — Urology, St. Joseph's Hospital, University of Western Ontario
Locations (6):
- Canada (6):
  - Alberta Urology Institute Research Centre, Edmonton, Alberta
  - Prostate Centre at Vancouver General Hospital, Vancouver, British Columbia
  - Can-Med Clinical Research Inc, Victoria, British Columbia
  - Hamilton District Urology Associaton, Hamilton, Ontario
  - Centre for Advanced Urological Research at Queen's University, Kingston, Ontario
  - Urology Clinic & Prostate Centre, St. Joseph's Hospital, St. Joseph's Health Care London, London, Ontario